CLINICAL TRIAL: NCT00921661
Title: A Dose-escalation Study of the Safety, Tolerability, and Pharmacokinetics of Intravenous Aflibercept in Combination With Intravenous Irinotecan/5-fluorouracil/Isovorin (FOLFIRI) Administered Every 2 Weeks in Patients With Metastatic Colorectal Cancer
Brief Title: Study of Intravenous Aflibercept in Combination With FOLFIRI in Japanese Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD10794
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Colorectal Neoplasms; Neoplasm Metastasis
Keywords: oxaliplatin; 5-FU; Folinic Acid
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AVE0005 (aflibercept) (Experimental)
  Interventions: Drug: AVE0005 (aflibercept)

INTERVENTIONS:
Drug: AVE0005 (aflibercept) — IV infusion

SUMMARY:
The primary objective is to determine the dose of aflibercept to be further studied in combination with irinotecan/5-fluorouracil/isovorin (FOLFIRI) in Japanese patients with metastatic colorectal cancer.

Secondary objectives of this study are to assess the safety profile of aflibercept, to determine the pharmacokinetics of aflibercept, to make a preliminary assessment of antitumor effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically proven malignant tumor of the colon or rectum which is metastatic and inoperable.
* Patients must have received at least one prior line of treatment with any standard of care, who have failed the treatment, or who have not been eligible for standard of care for safety reasons.

Exclusion Criteria:

* Treatment with chemotherapy, hormone therapy, radiotherapy, surgery, blood products, or any investigational agent within 28 days.
* ECOG Performance Status>1
* Anticipated need for a major surgical procedure or radiation therapy during the study.
* Uncontrolled malignant ascites.
* History of brain metastases, spinal cord compression, or carcinomatous meningitis or new evidence of brain or leptomeningeal disease on screening CT or MRI scan.
* Pregnant or breast-feeding women.
* Uncontrolled hypertension
* Patients who have previously been treated with aflibercept
* History of abdominal fistula, GI perforation, or intra-abdominal abscess within the past 28 days.
* History of hypersensitivity to any recombinant proteins, irinotecan, fluoropyrimidine or isovorin.
* Known dihydropyrimidine dehydrogenase deficiency.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) combination with FOLFIRI | During the first 2 cycles (4 weeks) of study treatment

SECONDARY OUTCOMES:
physical examination, laboratory safety tests, adverse events | up to 60 days after last treatment
Pharmacokinetics | up to 90 days after last treatment
Tumor burden, endogenous free VEGF | every 3 cycles
Immunogenicity | up to 90 days after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Tokyo, Japan

REFERENCES:
- [Derived] Yoshino T, Yamazaki K, Yamaguchi K, Doi T, Boku N, Machida N, Onozawa Y, Asayama M, Fujino T, Ohtsu A. A phase I study of intravenous aflibercept with FOLFIRI in Japanese patients with previously treated metastatic colorectal cancer. Invest New Drugs. 2013 Aug;31(4):910-7. doi: 10.1007/s10637-012-9895-6. Epub 2012 Nov 20. PMID 23179335